CLINICAL TRIAL: NCT04395781
Title: Pediatric Acute and Critical Care COVID-19 Registry of Asia
Acronym: PACCOVRA
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: King Chulalongkorn Memorial Hospital (Other); Ramathibodi Hospital (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); Rumah Sakit Anak dan Bunda Harapan Kita (Unknown); National University Hospital, Singapore (Other); St. Marianna University School of Medicine (Other); Tokyo Metropolitan Children's Medical Center, Japan (Unknown); Aichi Children's Health and Medical Center, Japan (Unknown); RS H Adam Malik (Other); Children's Hospital of Chongqing Medical University (Other); Zhengzhou Children's Hospital, China (Other); Universiti Kebangsaan Malaysia Medical Centre (Other); Penang Hospital, Malaysia (Other Government); Vicente Sotto Memorial Medical Center (Unknown); Hyogo Prefectural Kobe Children's Hospital (Other); Singapore Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/2094
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: COVID; Pediatric Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Biospecimen Retention: Samples With DNA — Blood Respiratory fluid Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control cases: Children who suspected COVID-19 cases but tested negative for COVID-19
- Confirmed cases: Children who tested positive for COVID-19

SUMMARY:
In December 2019, an outbreak of pneumonia of unknown aetiology was first reported in the city of Wuhan, Hubei Province, People's Republic of China. Since then, a novel coronavirus, 2019 novel Coronavirus (2019-nCoV) has emerged as the most likely causative agent. To date, it has evolved into a pandemic involving over a million cases and thousands of deaths have been identified, including a high burden in countries like Italy, Spain, United Kingdom and the United States. This study aims to investigate the clinical epidemiology of 2019-novel coronavirus (2019-nCoV) pandemic in Asia.

DETAILED DESCRIPTION:
A retrospective/prospective outbreak study of all suspect cases admitted to hospital since the beginning of the pandemic (December 2019). Clinical and epidemiological information will be extracted from medical databases for analysis.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 suspected cases (by whatever definition)
* COVID-19 confirmed cases (based on PCR or serum specific IgM and IgG antibody of novel coronavirus; serum specific IgG of novel coronavirus from negative to positive or 4 times higher in convalescence than in acute phase)
* </=21years of age

Exclusion Criteria:

* COVID-19 suspected cases should not be SARSCoV-2

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children presenting to acute care hospitals within the PACCMAN collaborative sites.
Sampling Method: Non-Probability Sample
Enrollment: 1756 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-09 (Actual)

PRIMARY OUTCOMES:
Overall severity of illness | 60days (or duration of hospital stay)
  Mild, moderate, severe, critical

SECONDARY OUTCOMES:
Respiratory complications | 60days (or duration of hospital stay)
  e.g. URTI, bronchiolitis, pneumonia, pneumothorax, effusion, pneumonitis, ARDS
Respiratory support | 60days (or duration of hospital stay)
  e.g. oxygen, HFNC, NIV, mechanical ventilation
Other systems complications | 60days (or duration of hospital stay)
  e.g. cardiovascular, renal, hepatic, neurological, haematological dysfunction
Mortality | 60days (or duration of hospital stay)
Length of hospital stay | 60days (or duration of hospital stay)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ju Ming Wong, Principal Investigator — KK Women's and Children's Hospital
Locations (14):
- China (2):
  - Chongqing Hospital Children's Medical Center, Chongqing
  - Zhengzhou Children's hospital, Zhengzhou
- Post Graduate Institute of Medical Education and Research, Chandigarh, India
- Indonesia (2):
  - General Hospital H. Adam Malik, Medan
  - Murni Teguh Memorial Hospital, Medan
- St. Marianna University School of Medicine, Kanagawa, Japan
- Malaysia (5):
  - Universiti Kebangsaan Malaysia Medical Centre, Bandar Tun Razak, Kuala Lumpur
  - Hospital Enche' Besar Hajjah Khalsom, Kluang
  - University Malaya Medical Centre, Kuala Lumpur
  - Penang General Hospital, Pulau Pinang
  - Hospital Tuanku Ja'afar, Seremban, Malaysia, Seremban
- Aga Khan University Hospital, Karachi, Pakistan
- Singapore (2):
  - KK Women's and Children's Hospital, Singapore
  - National University Hospital, Singapore, Singapore